CLINICAL TRIAL: NCT02752685
Title: Phase II Study of Pembrolizumab and Nab-paclitaxel in HER-2 Negative Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-00441
Record Dates: First submitted 2016-04-25; First posted 2016-04-27 (Estimated); Results first posted 2024-03-06 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: Nab-Paclitaxel; Abraxane; MK-3475
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- HR-Positive Participants (Experimental): Participants with HR-positive metastatic breast cancer will receive nab-paclitaxel 100 mg/m2 on days 1 and 8 of the first 21-day treatment cycle. On the second 21-day treatment cycle, the participants will receive pembrolizumab 200 mg IV on the first day of the cycle, in addition to nab-paclitaxel 100 mg/m2 on days 1 and 8 of the cycle.
  Interventions: Drug: Pembrolizumab; Drug: Nab-Paclitaxel
- cTNBC Participants (Experimental): Participants with TNBC-positive metastatic breast cancer who in the chemotherapy run-in group (cNTBC) will receive nab-paclitaxel 100 mg/m2 on days 1 and 8 of the first 21-day cycle. On the second 21-day treatment cycle, the participants will receive pembrolizumab 200 mg IV on the first day of the cycle, in addition to nab-paclitaxel 100 mg/m2 on days 1 and 8 of the cycle.
  Interventions: Drug: Pembrolizumab; Drug: Nab-Paclitaxel
- iTNBC Participants (Experimental): Participants with TNBC-positive metastatic breast cancer in the immunotherapy run-in group (cNTBC) will receive pembrolizumab 200mg IV on day 1 of the first 21-day treatment cycle. nab-paclitaxel 100 mg/m2 on days 1 and 8 of the first 21-day cycle. On the second 21-day cycle, the participants will receive nab-paclitaxel 100 mg/m2 on days 1 and 8 of the cycle, in addition to pembrolizumab 200mg IV on day 1 of the cycle.
  Interventions: Drug: Pembrolizumab; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab
  Other Names: MK-3475
Drug: Nab-Paclitaxel
  Other Names: Abraxane

SUMMARY:
This is a single-arm open-label multi-cohort Phase II study evaluating the safety/tolerability and clinical activity of the combination of nab-paclitaxel and the antibody against programmed cell death 1 (PD-1), pembrolizumab, in patients with human epidermal growth factor receptor (HER-2) negative metastatic breast cancer (n=50). There will be two cohorts of patients consisting of a triple negative breast cancer (TNBC) cohort with 30 subjects and a hormone receptor (HR)-positive cohort with 20 subjects. There will be an initial safety run-in with 12 subjects from the TNBC and HR-positive cohort (~ 6 patients from each cohort). If no unexpected toxicity is observed (as defined in the study protocol), then enrollment will continue to complete both cohorts (30 total TNBC, 20 total in HR positive cohort). The subjects from the run in safety part will be included in the Phase II analysis. Tumor expression of programmed cell death ligand 1 (PD-L1) is not required for enrollment in the study, but will be assessed as possible predictive marker.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed adenocarcinoma of the breast that is either TNBC or HR positive/HER-2 negative. TNBC is defined as: ER/PR <1% and HER-2 negative disease (IHC 0-1+ or 2+ with HER2/17 ratio on FISH ≤1.8) according to ASCO/CAP guidelines11,67. HR positive is defined as: ER/PR >= 1% and HER-2 negative as per ASCO/CAP guidelines.
* Have received 0-2 lines of cytotoxic chemotherapy for metastatic breast cancer endocrine therapy and/or targeted therapy is allowed.
* Be willing and able to provide written informed consent/assent for the trial
* Be 18 years of age on day of signing informed consent.
* Have measurable disease based on RECIST 1.1.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the PI or designee.
* Have a performance status of 0 or 1 on the ECOG Performance Scale. Be willing to undergo tissue biopsies as mandatory as per protocol for patients with biopsy accessible disease.
* Must have </= Grade 1 pre-existing peripheral neuropathy (as per CTCAE).
* Demonstrate adequate organ function as defined in all screening labs should be performed within 10 days of treatment initiation.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. This applies even if the subject practices true abstinence* from heterosexual contact. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* A female subject of childbearing potential is a sexually mature women who (1) has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or (2) has not been naturally postmenopausal for at least 24 consecutive months [i.e., has had menses at any time during the preceding 24 consecutive months]. The female subject must: either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis), or agree to use, and be able to comply with, effective contraception without interruption (2 methods of birth control), 28 days prior to starting IP therapy (including dose interruptions), and while on study medication or for a longer period if required by local regulations following the last dose of IP.
* Male subjects must practice true abstinence* or agree to use a condom during sexual contact with a pregnant female or female of childbearing potential starting with the first dose of study therapy, during dose interruptions, and for up to 6 months following last dose of study therapy, even if he has undergone a successful vasectomy.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis).
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Taxane therapy within the past 3 months (90 days) prior to study Day 1.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that progressed or required treatment within the last five years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of/active pneumonitis requiring treatment with steroids or history of/active interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies, testing not mandatory).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2016-06; Primary Completion 2022-12-29 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Klar, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Perlmutter Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- HR-Positive Participants: Participants with HR-positive metastatic breast cancer will receive nab-paclitaxel 100 mg/m2 on days 1 and 8 of the first 21-day treatment cycle. On the second 21-day treatment cycle, the participants will receive pembrolizumab 200 mg IV on the first day of the cycle, in addition to nab-paclitaxel 100 mg/m2 on days 1 and 8 of the cycle.
  Pembrolizumab
  Nab-Paclitaxel
- cTNBC Participants: Participants with TNBC-positive metastatic breast cancer who in the chemotherapy run-in group (cNTBC) will receive nab-paclitaxel 100 mg/m2 on days 1 and 8 of the first 21-day cycle. On the second 21-day treatment cycle, the participants will receive pembrolizumab 200 mg IV on the first day of the cycle, in addition to nab-paclitaxel 100 mg/m2 on days 1 and 8 of the cycle.
  Pembrolizumab
  Nab-Paclitaxel
- iTNBC Participants: Participants with TNBC-positive metastatic breast cancer in the immunotherapy run-in group (cNTBC) will receive pembrolizumab 200mg IV on day 1 of the first 21-day treatment cycle. nab-paclitaxel 100 mg/m2 on days 1 and 8 of the first 21-day cycle. On the second 21-day cycle, the participants will receive nab-paclitaxel 100 mg/m2 on days 1 and 8 of the cycle, in addition to pembrolizumab 200mg IV on day 1 of the cycle.
  Pembrolizumab
  Nab-Paclitaxel
Period: Overall Study
Arm/Group | HR-Positive Participants | cTNBC Participants | iTNBC Participants
Started | 20 | 30 | 20
Completed | 19 | 29 | 19
Not Completed | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HR-Positive Participants | cTNBC Participants | iTNBC Participants | Total
Number analyzed (Participants) | 20 | 30 | 20 | 70
Age, Continuous [Median (Full Range); unit: years] | 56 [34 to 75] | 53 [33 to 74] | 55 [22 to 84] | 55 [22 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 30 | 20 | 70
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 | 7
  Not Hispanic or Latino | 18 | 28 | 17 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 5 | 7 | 13
  White | 15 | 19 | 7 | 41
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 20 | 30 | 20 | 70

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Best Overall Response Rate (BORR) of Complete Response or Partial Response
Description: Overall response measured by RECIST version 1.1 and will be used in this study for assessment of tumor response. Complete response (CR) defined as disappearance of all target lesions; and partial response (PR) defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to Year 2
Measure: Count of Participants; unit: Participants
Groups:
- iTNBC Participants: Participants with TNBC-positive metastatic breast cancer in the immunotherapy run-in group (iNTBC) will receive pembrolizumab 200mg IV on day 1 of the first 21-day treatment cycle. nab-paclitaxel 100 mg/m2 on days 1 and 8 of the first 21-day cycle. On the second 21-day cycle, the participants will receive nab-paclitaxel 100 mg/m2 on days 1 and 8 of the cycle, in addition to pembrolizumab 200mg IV on day 1 of the cycle.
  Pembrolizumab
  Nab-Paclitaxel
Arm/Group | HR-Positive Participants | cTNBC Participants | iTNBC Participants
Number analyzed (Participants) | 19 | 29 | 19
Participants | 5 | 9 | 10

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS defined as the time from initial treatment to documented disease progression or death.
Time Frame: Up to Year 2
Reporting Status: Not Posted, anticipated posting 2025-06

3. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from initial treatment to death due to any cause.
Time Frame: Up to Year 2
Reporting Status: Not Posted, anticipated posting 2025-06

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Percentage of patients whose disease shrinks or remains stable over a certain time period.
Time Frame: Up to Year 2
Reporting Status: Not Posted, anticipated posting 2025-06

5. Secondary Outcome: Duration of Response (DOR)
Description: Defined as the time from onset of response to progression or death due to any reason, whichever occurs earlier.
Time Frame: Up to Year 2
Reporting Status: Not Posted, anticipated posting 2025-06

ADVERSE EVENTS:
Time Frame: 2 years
Description: Systematic,- PI to monitor for AEs at every cycle visit. Note that Serious Adverse Event and All-Cause Mortality data are still being analyzed and will be provided once available.
Arm/Group | HR-Positive Participants | cTNBC Participants | iTNBC Participants
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/30 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/30 | 0/20
Other Adverse Events (participants affected / at risk) | 20/20 | 30/30 | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HR-Positive Participants (N=20) | cTNBC Participants (N=30) | iTNBC Participants (N=20)
Abdominal pain (Gastrointestinal disorders) | 4 | 6 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 8 | 10 | 10
Alkaline phosphatase increased (Investigations) | 5 | 3 | 11
Allergic reaction (Immune system disorders) | 1 | 0 | 0
Alopecia (Immune system disorders) | 10 | 10 | 3
Anemia (Blood and lymphatic system disorders) | 10 | 10 | 18
Anorexia (Metabolism and nutrition disorders) | 3 | 6 | 2
Anxiety (Psychiatric disorders) | 1 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 8 | 13 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 7 | 4
Bloating (Gastrointestinal disorders) | 2 | 1 | 1
Thrombocytopenia (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 2 | 1
Blurred vision (Eye disorders) | 2 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 3 | 3
Chills (General disorders) | 4 | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 6 | 8 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 11 | 6
Creatinine increased (Investigations) | 4 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 3 | 2
Diarrhea (Gastrointestinal disorders) | 8 | 9 | 7
Dizziness (Nervous system disorders) | 3 | 3 | 4
Dry eye (Eye disorders) | 1 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Dysgeusia (Nervous system disorders) | 3 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 11 | 8
Ear and labyrinth disorder (Ear and labyrinth disorders) | 1 | 0 | 0
Edema limbs (General disorders) | 1 | 1 | 1
Increased LDH (Endocrine disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Esophageal pain (Gastrointestinal disorders) | 1 | 0 | 0
Eye Infection (Eye disorders) | 1 | 0 | 0
Light Flash (Eye disorders) | 1 | 0 | 0
Vision Change (Eye disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 1
Fatigue (General disorders) | 8 | 12 | 9
Fever (General disorders) | 6 | 6 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Flu like symptoms (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Gait disturbance (General disorders) | 1 | 1 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 4
Esophageal Spams (Gastrointestinal disorders) | 1 | 0 | 0
Oral Swelling (Jaw/Gum) (Gastrointestinal disorders) | 1 | 0 | 0
Early Satiety (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Mouth Sores) (Gastrointestinal disorders) | 1 | 1 | 1
Lip Mouth Sores Right Buccal, Tongue (Gastrointestinal disorders) | 1 | 0 | 0
Biopsy Site Pain (General disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 5 | 7 | 6
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hot flashes (Vascular disorders) | 2 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1 | 5
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2 | 5
Hyponatremia (Metabolism and nutrition disorders) | 4 | 3 | 6
Hypotension (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypothyroidism (Endocrine disorders) | 4 | 3 | 2
Seasonal allergies (Immune system disorders) | 1 | 3 | 0
chest discomfort- upper respiratory infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 1 | 3 | 0
Chest discomfort-UTI (Infections and infestations) | 1 | 0 | 0
chest discomfort-Periocular/Orbital Rash Bilateral (Infections and infestations) | 1 | 0 | 0
chest discomfort-viral gastroenteritis (Infections and infestations) | 1 | 0 | 0
chest discomfort-Oral Thrush (Infections and infestations) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 5 | 3
Irregular menstruation (Reproductive system and breast disorders) | 1 | 0 | 0
Lip infection (Infections and infestations) | 1 | 1 | 0
Localized edema (Vascular disorders) | 2 | 3 | 5
Lymphedema (Vascular disorders) | 2 | 3 | 2
Mucositis oral (Gastrointestinal disorders) | 2 | 2 | 1
joint stiffness-left fingers (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Leg Cramps (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Aching Feet (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 3
Nausea (Gastrointestinal disorders) | 12 | 13 | 13
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Aggitation (Nervous system disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 3 | 8 | 4
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 1 | 0
Pain (Gastrointestinal disorders) | 13 | 12 | 8
Palpitations (Cardiac disorders) | 1 | 5 | 1
Papulopustular rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Paresthesia (Musculoskeletal and connective tissue disorders) | 4 | 6 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Periorbital edema (Eye disorders) | 1 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 6 | 8
Platelet count decreased (Investigations) | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 6 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 6 | 6
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
hesitancy (Renal and urinary disorders) | 1 | 0 | 0
dysuria (Renal and urinary disorders) | 1 | 0 | 0
Vaginal Irritation Desquamation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Scalp Folliculitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Erythema (Mediport Site) (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Contrast Initiated Right Hand Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritic Rash - Upper Chest (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythematous Patches AC + Popliteal Fossa (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Left Foot Bottom Skin Peeling (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Soft Tissue Lump (Left Flank) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 3 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 3
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 2 | 3 | 1
Urinary frequency (Renal and urinary disorders) | 5 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 5 | 1
Urinary tract obstruction (Renal and urinary disorders) | 5 | 0 | 0
Vaginal dryness (Reproductive system and breast disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 8 | 8 | 4
Weight gain (Investigations) | 1 | 0 | 0
Weight loss (Investigations) | 1 | 2 | 0
White blood cell decreased (Investigations) | 1 | 1 | 2
Wound infection (Infections and infestations) | 1 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Edema face (General disorders) | 0 | 1 | 1
decreased T4 Free (Endocrine disorders) | 0 | 1 | 0
increased TSH (Endocrine disorders) | 0 | 1 | 0
T3 Increased (Endocrine disorders) | 0 | 1 | 0
T4 Increased (Endocrine disorders) | 0 | 1 | 0
TSH decreased (Endocrine disorders) | 0 | 1 | 0
decreased visual activity (when reading small print) (Eye disorders) | 0 | 1 | 0
Right upper eye swelling (Eye disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 1 | 0
Facial pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Floaters (Eye disorders) | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
blood on toilet tissue (Gastrointestinal disorders) | 0 | 1 | 0
gas (Gastrointestinal disorders) | 0 | 1 | 0
loose stool (Gastrointestinal disorders) | 0 | 1 | 0
Ulcers (Gastrointestinal disorders) | 0 | 1 | 0
Lower leg extremity edema (Gastrointestinal disorders) | 0 | 1 | 0
left hand edema (Gastrointestinal disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 1 | 2
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 5
Hypertension (Vascular disorders) | 0 | 2 | 0
Influenza A (Infections and infestations) | 0 | 1 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0
possible device related infection (Infections and infestations) | 0 | 1 | 0
Rhinovirus (Infections and infestations) | 0 | 1 | 0
sinus infection (Infections and infestations) | 0 | 1 | 0
Left Ankle Sprained (Injury, poisoning and procedural complications) | 0 | 2 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 5
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Baker's cyst L.popliteal fossa (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Baker's cyst right leg (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Feet Soreness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Left Toes Cramping (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Right Toes Cramping (Curling) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Nail infection (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 3 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Right Breast Feeling Swollen (Reproductive system and breast disorders) | 0 | 1 | 0
Spotting (Reproductive system and breast disorders) | 0 | 1 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Bilateral Redness of Feet (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Chest induration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ecchymosis Right Heel (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Ingrown Toe Nails (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Left Breast Burning Sensation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Lesion on Right Chest (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Lipoma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
LLE erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Neck Rash - Left Trapezium (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
onycholysis loose nails (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
right breast/chest erythema (dermatitis) (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Tinea Capitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Verrusa Vulgaris (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 2 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 2 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 1 | 0
Vulval infection (Reproductive system and breast disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Albumin (Blood and lymphatic system disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Breast infection (Infections and infestations) | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cardiac troponin I increased (Investigations) | 0 | 0 | 2
Cardiac troponin T increased (Investigations) | 0 | 0 | 1
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 1
Confusion (Nervous system disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
DVT (Vascular disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Edema Cerebral Peritumoral (Nervous system disorders) | 0 | 0 | 1
Mouth Abrasions (Oral Mucosa) (Gastrointestinal disorders) | 0 | 0 | 1
Heart failure (Cardiac disorders) | 0 | 0 | 1
Hematoma (Vascular disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 3
Folic Acid Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 1
Pain- Lower Back (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain Right Breast (Reproductive system and breast disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Left Nipple Discharge (Reproductive system and breast disorders) | 0 | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Right neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Left Breast scarring (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Heat Rash Arms (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Facial acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash Right Nare (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
skin infection (Infections and infestations) | 0 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
tachycardia (Cardiac disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT02752685/Prot_SAP_000.pdf